CLINICAL TRIAL: NCT04421534
Title: Efficacy and Safety of Lactoferrin as an Adjunct Therapeutic Agent for COVID-19
Brief Title: Utility of Lactoferrin as an Adjunct Therapeutic Agent for COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gamal Esmat, Professor of Endemic Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUKA-001
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: COVID-19; lactoferrin
MeSH Terms: conditions — COVID-19 | interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care in addition to 400 mg lactoferrin (Experimental): Standard of care treatment; as per MOHP protocol, in addition to 400 mg oral lactoferrin daily [two sachets 100 mg granules (Pravotin sachets, Hygint, Egypt) in 1/4 glass of water twice a day before meals]
  Interventions: Drug: Lactoferrin
- Standard of care in addition to 600 mg lactoferrin (Experimental): Standard of care treatment; as per MOHP protocol, in addition to 600 mg oral lactoferrin daily [three sachets 100 mg granules (Pravotin sachets, Hygint, Egypt) in 1/4 glass of water twice a day before meals]
  Interventions: Drug: Lactoferrin
- Standard of care only (Active Comparator): Standard of care treatment; as per MOHP protocol
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin — adding lactoferrin to standard of care treatment regimens
  Other Names: Standard of care treatment regimens

SUMMARY:
There is currently no clinically proven specific antiviral agent available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, remains the most important management strategy.

Since its discovery, lactoferrin and its related peptides are mainly considered to be important non-specific host defense molecules against a broad range of viruses including SARS-CoV, which is closely related to SARS-CoV-2 that causes COVID-19. Lactoferrin has been found to experimentally inhibit viral entry in murine coronavirus, and human coronaviruses hCOV-NL63 and pseudotyped SARS-CoV. Besides reducing viral entry, lactoferrin can also suppress virus replication after the viral entry.

Another major aspect of lactoferrin bioactivity relates to its immunomodulatory and anti-inflammatory functions. Current thinking suggests that mortality from COVID-19 is not simply due to viral infection but is a result of a cytokine storm associated with hyper-inflammation leading to acute respiratory distress and subsequent mortality. A cytokine profile in severe COVID-19 cases is characterized by increases in cytokines and acute phase reactants and ferritin. In this regard, lactoferrin was demonstrated to reduce IL-6, TNF a, and downregulate ferritin in experimental settings simulating sepsis.

In this study, we aim to study the potential application of lactoferrin against SARS-CoV-2 and propose the possibility of using different doses of supplemental lactoferrin as a potential adjunct treatment for COVID-19.

DETAILED DESCRIPTION:
COVID-19 has a wide clinical spectrum ranging between asymptomatic infection, mild upper respiratory tract symptoms, and severe viral pneumonia that may result in respiratory failure and finally death. There is currently no clinically proven specific antiviral agent available for SARS-CoV-2 infection. Supportive treatment, including oxygen therapy, conservation fluid management, and broad-spectrum antibiotics to cover secondary bacterial infection, remains the most important management strategy.

Lactoferrin is a highly conserved pleiotropic iron-binding 80-kDa glycoprotein of the transferrin family that is expressed and secreted by glandular cells and found in most body fluids with especially high concentrations in mammalian milk. Since its discovery, lactoferrin and its related peptides are mainly considered to be important non-specific host defense molecules against a broad range of viruses including SARS-CoV, which is closely related to SARS-CoV-2 that causes COVID-19. Lactoferrin has been found to experimentally inhibit viral entry in murine coronavirus, and human coronaviruses hCOV-NL63 and pseudotyped SARS-CoV. Given the homology of SARS-CoV and SARS-CoV-2 spike protein structures, as well as both viruses depending on the same ACE2 receptor for cell entry, it is likely that lactoferrin can inhibit SARS-CoV-2 invasion as in the case of SARS-CoV. Besides reducing viral entry, lactoferrin can also suppress virus replication after the viral entry as in the case of HIV.

Another major aspect of lactoferrin bioactivity relates to its immunomodulatory and anti-inflammatory functions. Current thinking suggests that mortality from COVID-19 is not simply due to viral infection but is a result of a cytokine storm associated with hyper-inflammation leading to acute respiratory distress and subsequent mortality. A cytokine profile in severe COVID-19 cases is characterized by increases in cytokines and acute phase reactants such as interleukin IL-6, tumor necrosis factor-a (TNFa) and ferritin. In this regard, lactoferrin was demonstrated to reduce IL-6, TNF a, and downregulate ferritin in experimental settings simulating sepsis.

The aim of this study is to confirm the antiviral properties and immunomodulatory mechanisms of lactoferrin within the context of its potential application against SARS-CoV-2 and propose the possibility of supplemental lactoferrin in different doses as a potential adjunct treatment for COVID-19.

The clinical data as well as the demographic information will be collected from the clinicians involved in the project. All samples will be collected according to the approved research protocols. During this period, the database entry platforms will be formed.

Eligible patients will be randomly distributed in 3 groups:

Group 1 (n=50): standard of care treatment; as per Egyptian Ministry of Health and Population (MOHP) protocol, in addition to 400 mg oral lactoferrin daily Group 2 (n=50): standard of care treatment; as per MOHP protocol, in addition to 600 mg oral lactoferrin daily Group 3 (n=50): standard of care treatment; as per MOHP protocol (control group)

The trial will be done according to the principles of the Declaration of Helsinki and the Good Clinical Practice guidelines.

Patients will be assessed daily on a scale reflecting a range from uninfected to dead, where 0 is "no clinical or virological evidence of infection", 1 is "no limitation of activities", 2 is "limitation of activities", 3 is "hospitalized, no oxygen therapy", 4 is "oxygen by mask or nasal prongs", 5 is "non-invasive ventilation or high-flow oxygen", 6 is "intubation and mechanical ventilation", 7 is "ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)", and 8 is "death".

Serial oropharyngeal swab samples will be obtained after treatment until discharge or death had occurred.

ELIGIBILITY:
Inclusion Criteria:

* Positive reverse-transcriptase-polymerase chain- reaction (RT-PCR) assay for SARS- CoV-2 in a respiratory tract sample.

Exclusion Criteria:

* Known allergy or hypersensitivity to the used medications
* Severe symptoms: respiratory insufficiency that requires admission in intensive care unit or mechanical ventilation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | 28 days
  time from randomization to improvement of two points on used scale or live discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Rate of virological cure | 28 days
  time from randomization to cure (2 SARS-COV-2 PCR samples negative with 48 hours apart)